CLINICAL TRIAL: NCT02165202
Title: HPTN 076 - Phase II Safety and Acceptability of an Investigational Injectable Product, TMC278 LA, for Pre-Exposure Prophylaxis (PrEP)
Brief Title: Phase II Safety and Acceptability of an Investigational Injectable Product, TMC278LA, for Pre-Exposure Prophylaxis
Acronym: TMC278LA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: HPTN 076; 1015131 (Other Grant/Funding Number: Bill & Melinda Gates Foundation (along with NIH for HPTN)); UM1AI068619 (NIH)
Record Dates: First submitted 2014-05-21; First posted 2014-06-17 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: HIV Pre-exposure Prophylaxis;; long-acting injectable;; HIV PrEP;; biomedical HIV prevention research
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rilpivirine (Active Comparator): Arm 1: Participants randomized to the active arm will receive rilpivirine 25 mg capsules once daily for four weeks to be taken orally with a meal. Participants will then receive IM injections of TMC278 LA, 1200 mg dose, at eight week intervals (at Weeks 4, 12, 20, 28, 36 and 44). On each dosing occasion 1200 mg of TMC278 LA will be delivered in two, 2 mL injections, one in each gluteus maximus muscle. All participants will receive a total of six doses (12 IM injections).
  Interventions: Drug: Rilpivirine
- Placebo (Placebo Comparator): Arm 2: Participants randomized to the placebo arm will receive placebo capsules once daily for four weeks to be taken orally with a meal. Participants will then receive IM injections of saline (0.9% NaCI) at eight week intervals (at Weeks 4, 12, 20, 28, 36 and 44). On each dosing occasion placebo will be delivered in two, 2 mL injections, one in each gluteus maximus muscle. All participants will receive a total of six doses (12 IM injections).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilpivirine — Rilpivirine (TMC278), a non-nucleoside reverse transcriptase inhibitor (NNRTI) is a substituted diaryl-pyrimidine (DAPY) derivative with potent antiviral activity against HIV. It is approved by the US FDA for once daily oral administration and is effective as part of treatment for ARV-na'ive HIV-infected patients as rilpivirine 25 mg capsules. It is also co-formulated with TDF and FTC for use as a once- daily single fixed-dose combination (Complera™).
  Arms: Rilpivirine
Drug: Placebo — Participants randomized to the placebo arm will receive oral placebo capsules prior to injection of saline solution (0.9%NaCI). Participants will be observed while taking the study product by site staff on approximately six occasions during the first two weeks of the oral run-in at Week 0 (Enrollment), at Week 2 (Oral Run-in Safety Visit), and on four separate DOT visits between Weeks 0 and 2. Cervicovaginal and rectal fluid will be collected for PK studies at a single follow-up visit.
  Arms: Placebo

SUMMARY:
This is a multi-site, double-blinded, two-arm, two:one, randomized, trial comparing the safety of an intramuscular (IM) injection of TMC278 LA to a placebo given once every eight weeks over a 40 week period among sexually active, HIV- uninfected women.

DETAILED DESCRIPTION:
This is a multi-site, double-blinded, two-arm, two:one randomized, placebo-controlled trial comparing the safety of TMC278 LA for 48 weeks after the initial 1M injection to a saline (0.9%NaCI) placebo IM injection among sexually active, HIV-uninfected women who are assessed by the clinic staff as being at "low risk" for HIV acquisition (in keeping with a safety trial). Approximately 132 women will be randomized to TMC278 LA and placebo in approximately a two:one ratio (88 and 44 in the TMC278 LA and placebo arm, respectively).

Approximately 96 women will be enrolled in SSA and approximately 36 women will be enrolled in the US. In order to screen for initial safety and tolerability of the active product, a run-in period with oral rilpivirine will precede the injection of TMC278 LA. Participants randomized to the placebo arm will receive oral placebo capsules prior to injection of saline solution (0.9%NaCI). Participants will be observed while taking the study product by site staff on approximately six occasions during the first two weeks of the oral run-in at Week 0 (Enrollment), at Week 2 (Oral Run-in Safety Visit), and on four separate DOT visits between Weeks 0 and 2. Cervicovaginal and rectal fluid will be collected for PK studies at a single follow-up visit. A subset of approximately 24 women at US sites will have vaginal tissue collection for PK studies at a single follow-up visit (Tissue Subset).

Participants who present with Grade 2 or greater RELATED AEs during the oral-run in phase will not receive the injectable TMC278 LA. Participants who present with Grade 3 or 4 UNRELATED AEs will not proceed to the injectable phase unless approved by the Clinical Management Committee (CMC).

Arm 1: Participants randomized to the active arm will receive rilpivirine 25 mg capsules once daily for four weeks to be taken orally with a meal. Participants will then receive IM injections of TMC278 LA, 1200 mg dose, at eight week intervals (at Weeks 4, 12, 20, 28, 36 and 44). On each dosing occasion 1200 mg of TMC278 LA will be delivered in two, 2 mL injections, one in each gluteus maximus muscle. All participants will receive a total of six doses (12 IM injections).

Arm 2: Participants randomized to the placebo arm will receive placebo capsules once daily for four weeks to be taken orally with a meal. Participants will then receive IM injections of saline (0.9% NaCI) at eight week intervals (at Weeks 4, 12, 20, 28, 36 and 44). On each dosing occasion placebo will be delivered in two, 2 mL injections, one in each gluteus maximus muscle. All participants will receive a total of six doses (12 IM injections).

Study sites:

* Bronx Prevention Center CRS, USA
* New Jersey Medical School CRS, USA
* Emavundleni CRS, Cape Town, South Africa
* Spilhaus CRS, Harare, Zimbabwe

ELIGIBILITY:
Inclusion Criteria: Women who meet all of the following criteria will be eligible for inclusion in the study:

* Women, 18- 45 years (inclusive) of age at Enrollment
* Female at birth
* Willing and able to provide informed consent to take part in the study
* Willing and able to provide adequate locator information
* Willing and able to provide acceptability and adherence assessments throughout the study
* Understands and agrees to local reporting requirements for sexually transmitted infections (STis)
* No evidence of an active STI, women who have an STI (Chlamydia trachomatis (CT), Neisseria gonorrhoeae (GC), or syphilis) identified at the Screening visit are ineligible*
* Per participant report, no diagnosis of GC, CT, or syphilis in the last 6 months
* Availability to return for all study visits and participate in all study-related procedures, barring unforeseen circumstances
* Per participant report, using (or willing to use) an acceptable form of contraception (e.g., intrauterine device [IUD], hormonal contraception [DMPA], oral, injectable, transdermal patch, implants) from screening until one month after last study visit or surgical sterilization of the participant
* Must agree to use condoms for the duration of the study
* Must agree not to participate in other concurrent drug or vaccine trials
* Normal laboratory values**

(HIV tests performed at Screening and Enrollment are non- reactive/negative (see Study Specific Procedures (SSP) Manual)

* Hemoglobin (women) =:: 10.5 g/dL
* Absolute neutrophil count1,000 cells/mm 3
* Platelet count=:: 100,000/mm3
* Calculated creatinine clearance =:: 70 mL!minute using the Cockcroft-Gault equation
* Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) < 2 times the upper limit of normal (ULN)
* Total bilirubin < 2.5 ULN
* Urine protein< 2+

  * Women who have an STI identified at the Screening visit (CT, GC, or syphilis) will be provided treatment but are ineligible. Women who report having CT, GC, or syphilis in the last six months are ineligible.

    * Specimens for Screening labs must be obtained within 28 days prior to study Enrollment.

3.1.1 Inclusion Criteria for the Tissue Subset (US sites only) A subset of approximately 24 participants at US sites will participate in more intensive sampling of vaginal tissue during Week 36 (preferred) or Week 44.

For these participants, the following additional criteria need to be met:

•Satisfactory Pap results in the 12 calendar months prior to biopsy consistent with Grade 0 according to the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Version 1.0, December 2004 (Clarification dated August 2009), or satisfactory evaluation with no treatment required of Grade 1 or higher Pap result per American Society for Colposcopy and Cervical Pathology (ASCCP) guidelines in the 12 calendar months prior to biopsy is required, as indicated.

If there is no documentation of satisfactory Pap results, and if indicated, the participant should be offered to have the test performed by the site prior to enrollment in the Tissue Subset. If Pap testing is indicated and participants decline, they are not eligible for the Tissue Subset.

* In addition to documentation of satisfactory Pap results, women must have normal laboratory results for coagulation tests to be eligible for the Tissue Subset. Abnormal coagulation test results may indicate an increased risk of bleeding.
* Women have to be willing to abstain from vaginal intercourse and practices involving insertion of anything in the vagina (drug, douche, penis, or sex toy) for 3 days prior to vaginal biopsy and for 7 days post-biopsy, to minimize risk of HIV-1 infection and bleeding complications after the procedure.
* Participants must not be pregnant at the time of vaginal sampling, based on pregnancy test results from previous visits and on the result of urine pregnancy test performed on the same day before the proposed vaginal sampling.
* Women undergoing biopsy must have received all prior injections of study product, in accordance with the protocol, to be eligible for inclusion.

Exclusion Criteria: Women who meet any of the following criteria will be excluded from the study:

* Experiencing early menopause using clinical criteria (amenorrhea greater than six months in absence of pregnancy) or a prior report of an abnormal Follicle Stimulating Hormone (FSH) test
* PrEP or post-exposure prophylaxis (PEP) for HIV exposure within 90 days prior to Screening
* Pregnant or last pregnancy outcome 90 days or less prior to Screening
* Currently breastfeeding
* Intends to become pregnant during the period of study participation
* Experiencing uncontrolled depression or active suicidal ideation
* History of recurrent urticaria
* Any history of anaphylaxis or severe allergy resulting in angioedema
* Any serious acute, chronic, or progressive disease (e.g. known history of neoplasm, cancer, insulin-dependent diabetes, cardiac disease, auto-immune disease), or with signs of cardiac disease, renal failure, or severe malnutrition
* Any laboratory abnormalities that are Grade 2 or higher, according to the DAIDS Toxicology tables (please see Section 6.1 for a list of Screening laboratory tests)
* Recreational injection drug use in the 52 weeks prior to screening
* Participating or plans to participate in another research study involving study drugs, vaccines or medical devices
* Participated in another research study involving study drugs, vaccines or medical devices within the four weeks prior to screening; may be longer than four weeks depending on half-life of study drug
* Past participation in an HIV vaccine study
* Has plans to relocate and cannot attend the visits at the clinic
* Per participant report at Screening, current or anticipated ongoing use and/or unwillingness to abstain from contraindicated medications or supplements (listed in the SSP Manual)
* Abnormal resting EKG at screening including:
* Abnormal sinus rhythm (heart rate below 40 or above 100 beats per minute)
* QTcF interval> 450 ms
* QRS interval < 50 ms
* QRS interval > 120 ms
* PR interval> 210 ms
* History of additional risk factors for Torsade de Pointes (TdP), such as heart failure, hypokalemia, hypomagnesia, family history of known long QT syndrome, or sudden death at young age (S 40 years) in a first-degree relative (i.e., biological parent, sibling, or offspring)
* Currently active Tuberculosis (TB), or undergoing treatment for the same (by self-report)
* Any signs or symptoms consistent with acute (pre-seroconversion) HIV infection, or self-reported concern about recent HIV infection
* Any reactive or positive HIV test at Screening or Enrollment, even if the person is confirmed to be HIV-uninfected
* Has any other condition that, in the opinion of the site loR or designee, would preclude informed consent, make study participation unsafe, interfere with adherence, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives (e.g., at increased risk of cardiovascular vents)

Women who do not meet eligibility criteria because of an abnormal EKG, risk factors for TdP, an STI (GC, CT, or syphilis) present at Screening or report of an STI (GC, CT, or syphilis) in the past 6 months, or a history of arrhythmia may not be re-screened.

Women who present at Screening with symptoms consistent with an acute HIV infection or who have a reactive HIV test may not be re-screened. Women who do not meet eligibility criteria for the study for other reason(s) may be re-screened at a future date at the discretion of the site loR.

3.2.1 Exclusion Criteria for the Tissue Subset (US sites only)

Participants of the Tissue Subset must meet the above eligibility criteria to be enrolled in HPTN 076. Participants interested in participating in the Tissue Subset must meet additional inclusion and exclusion criteria. Women who meet any of the following criteria will be excluded from the Tissue Subset:

* Unwillingness to abstain from the following medications for a period of 10 days before a biopsy procedure:
* Aspirin*
* Non-steroidal anti-inflammatory drugs (NSAIDS)

  *Daily use of low-dose aspirin (no more than 81 mg) is allowed at the discretion of the loR.
* Unwillingness to abstain from the following medications for 3 days prior to vaginal biopsy and for 7 days post-biopsy: Heparin, including Lovenox®, Warfarin, Plavix® (clopidogrel bisulfate), and any other drugs that are associated with increased risk of bleeding following biopsy procedures at the discretion of the loR.
* Carcinoma in situ of the cervix or invasive cervical cancer. Abnormalities of the vaginal mucosa or significant vaginal symptom(s), which in the opinion of the loR represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, and infectious or inflammatory condition of the local mucosa).
* Hysterectomy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04-13 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Justman, MD, Principal Investigator — Bronx-Lebanon Hospital Center Clinical Research Site; Shobha Swaminathan, MD, Principal Investigator — New Jersey Medical School Clinical Research Site; Zvavahera Michael Chirenje, MD, MSc, Principal Investigator — Spilhaus Clinical Research Site; Linda-Gail Bekker, PhD, Study Chair — The Desmond Tutu HIV Centre
Locations (4):
- United States (2):
  - New Jersey Medical School Clinical Research Center, Newark, New Jersey
  - Bronx Prevention Center, The Bronx, New York
- Emavundleni Clinical Research Site, Cape Town, South Africa
- Spilhaus Clinical Research Site, Belgravia, Harare, Zimbabwe

REFERENCES:
- [Background] Bekker LG, Beyrer C, Quinn TC. Behavioral and biomedical combination strategies for HIV prevention. Cold Spring Harb Perspect Med. 2012 Aug 1;2(8):a007435. doi: 10.1101/cshperspect.a007435. PMID 22908192
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Soto RJ, Ghee AE, Nunez CA, Mayorga R, Tapia KA, Astete SG, Hughes JP, Buffardi AL, Holte SE, Holmes KK; Estudio Multicentrico Study Team. Sentinel surveillance of sexually transmitted infections/HIV and risk behaviors in vulnerable populations in 5 Central American countries. J Acquir Immune Defic Syndr. 2007 Sep 1;46(1):101-11. PMID 17972366
- [Background] Coates TJ, Richter L, Caceres C. Behavioural strategies to reduce HIV transmission: how to make them work better. Lancet. 2008 Aug 23;372(9639):669-84. doi: 10.1016/S0140-6736(08)60886-7. Epub 2008 Aug 5. PMID 18687459
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- [Background] Haberer JE, Kahane J, Kigozi I, Emenyonu N, Hunt P, Martin J, Bangsberg DR. Real-time adherence monitoring for HIV antiretroviral therapy. AIDS Behav. 2010 Dec;14(6):1340-6. doi: 10.1007/s10461-010-9799-4. PMID 20809380
- [Background] Kashuba AD, Patterson KB, Dumond JB, Cohen MS. Pre-exposure prophylaxis for HIV prevention: how to predict success. Lancet. 2012 Jun 30;379(9835):2409-2411. doi: 10.1016/S0140-6736(11)61852-7. Epub 2011 Dec 6. No abstract available. PMID 22153566
- [Derived] Seneviratne HK, Tillotson J, Lade JM, Bekker LG, Li S, Pathak S, Justman J, Mgodi N, Swaminathan S, Sista N, Farrior J, Richardson P, Hendrix CW, Bumpus NN. Metabolism of Long-Acting Rilpivirine After Intramuscular Injection: HIV Prevention Trials Network Study 076 (HPTN 076). AIDS Res Hum Retroviruses. 2021 Mar;37(3):173-183. doi: 10.1089/AID.2020.0155. Epub 2021 Jan 13. PMID 33191765
- [Derived] Tolley EE, Li S, Zangeneh SZ, Atujuna M, Musara P, Justman J, Pathak S, Bekker LG, Swaminathan S, Stanton J, Farrior J, Sista N. Acceptability of a long-acting injectable HIV prevention product among US and African women: findings from a phase 2 clinical Trial (HPTN 076). J Int AIDS Soc. 2019 Oct;22(10):e25408. doi: 10.1002/jia2.25408. PMID 31651098

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants will be randomized to either the active product regimen or the placebo arm at enrollment. Participants randomized to active and placebo product will first be prescribed oral TMC278 (rilpivirine) 25 mg capsule and oral placebo capsule, once daily for four weeks as an oral run-in and then will receive IM injections at week 4.
Period: Oral Phase
Arm/Group | Rilpivirine | Placebo
Started | 91 (Participants Enrolled in the study) | 45 (Participants Enrolled in the study)
Completed (Participants who completed oral run in phase (0-week 4) and received at least 1 injection.) | 80 | 42
Not Completed | 11 | 3
Not completed — Refused further participation | 5 | 1
Not completed — Study product Related Toxicity | 1 | 0
Not completed — Unable to contact Participant | 1 | 1
Not completed — Clinical reasons | 1 | 0
Not completed — QTcF>500 ms or increase of>60 ms | 1 | 0
Not completed — CMC advised termination | 1 | 0
Not completed — Relocated, no follow-up planned | 1 | 0
Not completed — Abnormal EKG | 0 | 1
Period: Injection Phase
Arm/Group | Rilpivirine | Placebo
Started | 80 (Participants who received at least one injection.) | 42 (Participants who received at least one injection.)
Completed (Ppts who received at least 1 injection but were not discontinued or terminated till the end of study) | 70 | 36
Not Completed | 10 | 6
Not completed — Abnormal Lab Value | 5 | 1
Not completed — Reactive HIV or HIV Suspected | 0 | 2
Not completed — Unable to attend within Visit Window | 1 | 0
Not completed — QTcF>500 ms or increase of>60 ms | 0 | 1
Not completed — End of Study | 2 | 1
Not completed — Study Product related Toxicity | 1 | 0
Not completed — No longer interested | 0 | 1
Not completed — Participant unwilling to comply | 1 | 0

BASELINE CHARACTERISTICS:
Population: This template shows demographic characteristics of participants measured at Enrollment in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rilpivirine | Placebo | Total
Number analyzed (Participants) | 91 | 45 | 136
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [26 to 36] | 30 [25 to 39] | 31 [25 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 45 | 136
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 85 | 42 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 86 | 42 | 128
  White | 3 | 0 | 3
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 12 | 36
  Zimbabwe | 35 | 17 | 52
  South Africa | 32 | 16 | 48
Age, Categorical [Count of Participants; unit: Participants]
  18-25 | 22 | 14 | 36
  26-35 | 45 | 14 | 59
  36-45 | 24 | 17 | 41
Height [Median (Inter-Quartile Range); unit: cm] | 159 [153 to 165] | 158 [152 to 165] | 158 [153 to 165]
Weight [Median (Inter-Quartile Range); unit: kg] — Population: 1 participant was missing weight measurement
  kg
    number analyzed (Participants) | 90 | 45 | 135
    (all) | 76 [67 to 89] | 73 [63 to 88] | 75 [64 to 89]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Population: 1 participant was missing BMI
  kg/m^2
    number analyzed (Participants) | 90 | 45 | 135
    (all) | 31 [26 to 35] | 29 [27 to 35] | 30 [27 to 35]
Marital Status [Count of Participants; unit: Participants]
  Married/civil union/legal partnership | 45 | 18 | 63
  Living with primary or main partner | 5 | 2 | 7
  Have primary or main partner, not living | 15 | 6 | 21
  Single/divorced/widowed | 26 | 19 | 45
  Other | 0 | 0 | 0
Employment Status [Count of Participants; unit: Participants]
  Not employed | 60 | 22 | 82
  Part-time employment | 17 | 14 | 31
  Full-time employment | 14 | 9 | 23
Education [Count of Participants; unit: Participants]
  No schooling | 0 | 0 | 0
  Primary school, not complete | 16 | 11 | 27
  Primary school, complete | 58 | 27 | 85
  Secondary school, not complete | 7 | 3 | 10
  Secondary school, complete | 10 | 4 | 14
  Technical training, not complete | 0 | 0 | 0
  Technical training, complete | 0 | 0 | 0
  College or university, not complete | 0 | 0 | 0
  College or university, complete | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any Grade 2 or Higher AEs During Injection Phase
Description: Number of participants experiencing any Grade 2 or higher clinical and laboratory AEs to evaluate the safety of the injectable product, TMC278 LA (1200 mg dose administered at Weeks 4, 12, 20, 28, 36 and 44), through 48 weeks after initial injection (at Week 52) in women in SSA and the US.
Time Frame: Up to 52 weeks
Population: Participants who received at least one injection and were followed up to 52 weeks are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Rilpivirine | Placebo
Number analyzed (Participants) | 80 | 42
Participants | 59 | 31

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected from the time of enrollment to the end of the study. (From enrollment to week 76).
Description: Adverse Event data that were collected during injection phase from the time of first injection to week 52 are included in the Report showing list of other AEs excluding Serious AEs. (From week 4 to week 52).
Arm/Group | Rilpivirine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/91 | 0/45
Serious Adverse Events (participants affected / at risk) | 4/91 | 1/45
Other Adverse Events (participants affected / at risk) | 80/80 | 40/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilpivirine (N=91) | Placebo (N=45)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rilpivirine (N=80) | Placebo (N=42)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Induration (General disorders) | 5 (5) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 1 (1)
Injection site discharge (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 20 (20) | 1 (1)
Injection site granuloma (General disorders) | 4 (4) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 1 (1)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 6 (6) | 0 (0)
Injection site nodule (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 60 (60) | 17 (17)
Injection site pruritus (General disorders) | 29 (29) | 5 (5)
Injection site swelling (General disorders) | 29 (29) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 1 (1) | 2 (2)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 6 (6) | 3 (3)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary chlamydia infection (Infections and infestations) | 2 (2) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 2 (2)
Injection site abscess (Infections and infestations) | 1 (1) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 9 (9) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 6 (6)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 3 (3) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 3 (3) | 3 (3)
Vulvovaginitis trichomonal (Infections and infestations) | 3 (3) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 8 (8) | 2 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 29 (29) | 5 (5)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 17 (17) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 14 (14) | 5 (5)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Blood bicarbonate decreased (Investigations) | 11 (11) | 4 (4)
Blood bilirubin increased (Investigations) | 5 (5) | 5 (5)
Blood calcium decreased (Investigations) | 8 (8) | 6 (6)
Blood calcium increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 10 (10) | 4 (4)
Blood creatinine increased (Investigations) | 3 (3) | 3 (3)
Blood glucose decreased (Investigations) | 21 (21) | 6 (6)
Blood glucose increased (Investigations) | 19 (19) | 11 (11)
Blood phosphorus decreased (Investigations) | 16 (16) | 14 (14)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 3 (3) | 2 (2)
Body temperature increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram PR prolongation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 2 (2)
Haemoglobin decreased (Investigations) | 3 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1)
Platelet count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 8 (8) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (7)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 16 (16) | 11 (11)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (7) | 6 (6)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 21 (21) | 9 (9)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 5 (5) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No